CLINICAL TRIAL: NCT06089213
Title: Effects of Two Strategies for Preventing Falls in the Elderly Through Telerehabilitation: A Randomized Clinical Trial
Brief Title: Strategies for Preventing Falls in the Elderly
Acronym: Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Éder Kröeff Cardoso, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPSPoA
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Fall; Elderly; Prevention; Telehealth; Physical Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive services (Experimental): Otago exercises performed in "real-time" or "synchronous" mode of digital health care. It consists of direct communication between physiotherapist and the patient.
  Interventions: Other: real-time intervention
- Remote telemonitoring (Active Comparator): Otago exercises performed remotely, using technologies such as messaging apps. It consists of indirect communication between physiotherapist and the patient.
  Interventions: Other: real-time intervention

INTERVENTIONS:
Other: real-time intervention — An individual exercise program will be carried out at home, supervised remotely via videoconference.

SUMMARY:
Fall incidents are the third cause of chronic disability in the elderly, according to the World Health Organization (WHO). Recent reviews demonstrate that multifactorial and multicomponent intervention programs are effective in preventing falls in community-dwelling older adults. However, the application of these programs may not be accessible to a large part of the elderly population. The lack of continuity in the treatment of the consequences of falls, as well as the dissemination of prevention measures for this patient profile, could be minimized through the use of information and communication technologies. Method: This will be a randomized clinical trial that aims to evaluate the effects of two fall prevention strategies via telerehabilitation for elderly fallers after admission to an emergency room. It will be carried out by a multidisciplinary team with interventions for eight weeks and monitoring of outcomes over a period of four months. Patients will be evaluated regarding aspects of functionality in the second and month after the interventions and regarding the recurrence of falls during the four-month period. Discussion: The hypothesis is that the programs are viable in terms of accessibility to home training. However, to date, there is no evidence about the differences between these forms of interventions to prevent falls via telecare.

DETAILED DESCRIPTION:
To compare the effects of two different strategies for preventing falls through telerehabilitation for elderly fallers after admission to an emergency room.

ELIGIBILITY:
Inclusion Criteria:

* elderly fallers

Exclusion Criteria:

* neurological diseases

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Rate of Falls | four months
  After the intervention periods, participants will be followed for another 16 weeks. Every week, recurrences of falls will be recorded via telephone calls. You will be asked whether there were falls in the period

SECONDARY OUTCOMES:
Concern of falls | through study completion, an average of 1 year
  The assessment will consist of Self-efficacy tests for Falls
Balance | through study completion, an average of 1 year
  The assessment will consist of Timed-Up and Go test
Arms Muscle strength | through study completion, an average of 1 year
  Palm Grip Strength
Legs Muscle strength | through study completion, an average of 1 year
  Sitting and Rising from a Chair tests
Functionality | through study completion, an average of 1 year
  Katz Index on elderly functionality evaluation for the analysis of basic activities

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Pronto Socorro, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No